CLINICAL TRIAL: NCT05206175
Title: Demonstration of a Digital Care Program for Methamphetamine Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affect Therapeutics, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Methamphetamine Study; R43DA055394 (NIH)
Record Dates: First submitted 2021-12-27; First posted 2022-01-25 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Methamphetamine Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Arm (Experimental): Components of the Affect Therapeutic Program for MUD Components of the treatment services include: contingency management (CM; monetary incentives for drug tests negative for stimulants), the digital behavioral therapy curriculum (based on CBT) delivered via the Affect app on smartphones, weekly one-on-one telemedicine-based addiction counseling with clinical personnel, twice-weekly group therapy, and monthly psychiatrist appointments for evaluation and management and medication support, as needed.
  Interventions: Other: Affect Treatment Program for Methamphetamine Use Disorder

INTERVENTIONS:
Other: Affect Treatment Program for Methamphetamine Use Disorder — Telemedicine based group and individual therapy, drug screens, contingency management, therapeutic app engagement, psychiatric interventions for adjuvant medications.

SUMMARY:
This Phase I Small Business Innovation Research (SBIR) project will examine the technical merit and real-world feasibility of the Affect smartphone application ("app") as the core component of the Affect digital care program for treatment of methamphetamine use disorder (MUD).

DETAILED DESCRIPTION:
The project includes a clinical trial that will assemble data on the functionality of the app in engaging patients and delivering treatment components and related services, using outputs to guide rapid refinements of the app's functions (e.g., active and passive data collection, patient inference engine, triggers for clinician actions, user interfaces). The project will analyze these and other aspects of the app and program to assess their associations with patient engagement, participation, and retention, providing indication of the overall program's clinical utility.

Aim 1. Confirm the technical merit and feasibility of the Affect app and its delivery of the Affect digital care program in real-world practice based on results from the clinical trial.

Aim 2. Identify components of the Affect app and the Affect digital care program that correlate with patient engagement, participation, retention, and changes in methamphetamine use.

Aim 3. Use results to iteratively refine the Affect app and care program to improve treatment of MUD toward substantiating commercialization.

Demonstrating the technical merit, feasibility, and clinical utility of the Affect app and digital care platform could lead to improved clinical care for the 1.6 million people in the nation who need treatment for MUD. Results of this project have high potential to inform additional work to advance commercializability of the Affect program and its app, which would increase access to affordable, effective care for those who never receive treatment among the 2 million in need. If technical merit is demonstrated and the program is shown to be feasible and effective in retaining participants in treatment, the Affect app will be an important element in efficiently achieving optimum patient outcomes at reasonable cost.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, prospective participants must:

1. Be 18 years of age or older;
2. Have methamphetamine use disorder (MUD), confirmed by DSM-5 criteria for stimulant use disorder, methamphetamine type, endorsing >3 DSM-5 Checklist items (see Note below*);
3. Have stated interest in reducing and/or stopping methamphetamine use;
4. Have and be able to use a smartphone and agree to download and use the Affect app as part of study-related procedures;
5. Be English speaking and have reading capacity sufficient to understand explanations of study procedures and the informed consent to participate, which will be prepared at 7th-8th grade level;
6. Have a mailing address, P.O. box, or other means of receiving packages (for biologic sample kits) as a resident of Arizona;
7. Be able to freely give informed consent and be willing to electronically sign the digital informed consent to participate in the study;
8. Be willing to comply with study procedures, including use of the Affect app consistent with the study protocol and therapeutic activities.

   * Note: The inclusion criterion of MUD is established via the screening process involving questionnaires about meth use and the candidate's endorsement of DSM-5 criteria for MUD. We are confident in this process, given the fact that all of the participants (N=57) enrolled in our field study (Study # 1302084, IRB Tracking # 20210518, completed June 2021) tested positive for meth by the twice-weekly biologic tests during Weeks 1 and 2 of the intervention period, which confirms validity of the eligibility criterion of MUD determined by DSM-5 Checklist at screening.

Exclusion Criteria:

Individuals will be precluded from enrolling in the study if they endorse (or if there is indication of) any of the following items. Already-enrolled participants will be withdrawn from study participation upon emergence of an excluded condition (except pregnancy):

1. Serious medical condition (e.g., seizure, stroke, heart disease);
2. Serious mental illness (e.g., schizophrenia, bipolar, active suicidality);
3. Moderate- to severe-level opioid use disorder or alcohol use disorder at screening (DSM5 checklist);
4. Currently pregnant or planning on becoming pregnant (which may indicate a need for higher level of care to ensure safety of the woman and fetus);
5. Have been in a prior study of pharmacological or behavioral treatment for MUD within 6 months of study consent;
6. Be concurrently receiving behavioral or pharmacological services for treatment of MUD;
7. Have pending legal action or other situation that could inhibit consistent participation in the study or in study activities.
8. Have any other condition that, in the opinion of the PI and the Co-Investigator (Jeff DeFlavio, M.D.), would interfere with participation in and completion of this trial or would put individuals at risk to their well-being.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Participation retention and completion of treatment | Up to 8 weeks through the duration of treatment
  Participant retention and completion of the program will be measured as consistency of participant involvement through the end of the 8-week program, with criteria for completion being data on participation in >50% of potential therapeutic interactions and activities. A related "time in treatment" measure will also characterize retention (and detail aspects of engagement). At the end-of-program telephone interview, participants will be deemed to be either treatment completers (i.e., retained) or dropouts (not retained if out of program before the end of week 4 (excluding those who drop out in week 1).
Patient engagement and program adherence | Up to 8 weeks through the duration of treatment
  The nature/degree of participation in this study will be measured as the number of successfully "attended" therapeutic tasks/events/activities per the Affect app relative to not-attended events such as: scheduled/planned digital/virtual interactions for program activities (e.g., counseling, group meetings), completed biological assessments (remote drug biologic tests), and kept appointments with referred service providers (e.g., psychiatrists, physicians). Engagement with the Affect app components will be assessed via app-derived data on activity (i.e., duration, frequency, consistency of involvement with app-directed tasks). We will extract use-specific data on participants' interactions with the app, as well as results of surveys/questionnaires/focus groups to characterize associations of app and program components and procedures and their impacts on patient-level outcomes (e.g., retention in the program and meth use).
Effectiveness in reducing meth use | Through study completion, an average of 6 months
  The effectiveness outcome is determined by demonstrated reductions of meth use measured via a composite measure of self-reported meth use (daily Yes/No) plus results of biologic screens to provide indication of effectiveness. The criterion measure of clinically meaningful reduction of meth use will be 4 meth-negative biologic screens of the 8 possible biologic screens during the final 4 weeks of the 8-week program (concurring with self-report of no meth use).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Muhlner, Principal Investigator — Affect Therapeutics, Inc.
Locations (1):
- Affect Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT05206175/ICF_000.pdf